CLINICAL TRIAL: NCT00901420
Title: Comparison of Urodynamic Evaluation in Post-Radiation Salvage Prostatectomy Versus Prostatectomy-only Patients
Brief Title: Urodynamic Evaluation in Post-radiation Salvage Prostatectomy Patients
Status: Terminated | Type: Observational
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0384
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: Prostate; Urodynamic Evaluation; Prostatectomy; Salvage prostatectomy; Bladder compliance; Radiation Therapy; External beam radiation therapy; Quality-of-life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prostatectomy
  Interventions: Procedure: Urodynamics Test; Behavioral: Questionnaire
- Prostatectomy After Radiation Therapy
  Interventions: Procedure: Urodynamics Test; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Urodynamics Test — 90 Minute videotaped bladder function procedure involving pressure-monitoring catheters in bladder and rectum.
Behavioral: Questionnaire — Survey of urinary function and quality-of-life (regarding daily living after surgical treatment for prostate cancer), taking 30 minutes to complete.

SUMMARY:
Objectives:

The primary objective of this study is to determine whether bladder compliance is significantly lower in men who undergo prostatectomy for recurrence following primary radiation therapy than in men who undergo prostatectomy as primary treatment.

The secondary objective is to examine the quality-of-life items addressed in the UCLA Prostate Cancer Index for differences between the two populations. The investigators will also look at secondary objective urodynamic measures, such as bladder capacity, to assess for a difference.

DETAILED DESCRIPTION:
Study Participation:

You will come to the urology clinic for 1 visit. At this visit, a video urodynamics test will be performed. The urodynamics test is used to check bladder and urinary function using pressure and volume measurements with x-ray images.

Pressure-monitoring catheters will be inserted into your bladder and rectum, and your bladder function will be checked as the bladder is slowly filled with fluid. Measurements will then be made of your bladder capacity (the volume of urine the bladder can hold), bladder and abdominal (stomach) pressures, and bladder compliance (the bladder's ability to hold urine) throughout the course of this study. This procedure will take about 90 minutes to complete.

After the urodynamics test is completed, you will complete a questionnaire about your urinary function and your quality-of-life (regarding daily living after surgical treatment for prostate cancer). The questionnaire will take about 30 minutes to complete.

If you have had urodynamic testing with Dr. Westney within the past year, we would like your consent to use the data from that test, and also for completion of the questionnaire mentioned in the previous paragraph. You will complete this informed consent and questionnaire being sent with a return envelope and will not need to come to the urology clinic for a visit.

Length of Study:

Once you have completed the urodynamics testing and questionnaire, your participation on this study is complete.

This is an investigational study. The video urodynamics test is approved by the FDA and commercially available. Up to 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Men who have undergone radical prostatectomy, via an open or minimally invasive approach, as primary treatment for a diagnosis of prostate cancer.
2. Men who have undergone salvage prostatectomy for recurrence after first-line radiation therapy for prostate cancer.
3. Men who underwent prostatectomy at least one year prior to study entry date. Men who received perioperative (or peri-XRT) chemotherapy or hormone therapy are eligible.

Exclusion Criteria:

1. Men who underwent other primary or secondary treatments for prostate cancer--hormone therapy as only treatment, cryosurgery, adjuvant radiation after prostatectomy
2. Men with a history of neurogenic bladder, as demonstrated by previous urodynamics.
3. Men with a history of severe outlet obstruction due to longstanding benign prostatic hyperplasia. This will be demonstrated objectively by documentation in the patient's history of preoperative AUA symptom score greater than 15 or a history of urinary retention or nocturia greater than 2 episodes per night.
4. Men who underwent additional reconstructive procedures at the time of or subsequent to prostatectomy, including augmentation, urethral sling, or urinary diversion.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men, seen at MD Anderson Cancer Center, who underwent radical prostatectomy as the first-line treatment for their prostate cancer or underwent salvage prostatectomy for recurrence after first-line radiation treatment; or underwent prostatectomy at least one year prior to study entry date or received perioperative (or peri-XRT) chemotherapy or hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Comparison of Urodynamic Changes Related to Radiation Post Salvage Prostatectomy versus Prostatectomy Only | Compilation of patient urodynamics test completed in single 90 minute office visit
  Comparison of urodynamic changes related to radiation by performing urodynamics (measurement of bladder pressure, electrical activity, and radiographic imaging) in patients post salvage prostatectomy versus prostatectomy only, using a 2-sample t-test to test for differences between the 2 groups of men with respect to urodynamic score.

CONTACTS AND LOCATIONS:
Overall Officials: Ouida L. Westney, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org